CLINICAL TRIAL: NCT03249662
Title: Efficacy of Pain Management in Different Concentrations of Bupivacaine in Periarticular Injection and Plasma Concentrations of Bupivacaine in Patients Undergoing Bilateral Knee Arthroplasty
Brief Title: Efficacy of Pain Control in Different Bupivacaine Dose in Periarticular Injection in Bilateral Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: si111/2017
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Bilateral Total Knee Arthroplasty
Keywords: periarticular infiltration; postoperative pain management; plasma level of bupivacaine
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine 100 mg (Experimental): bupivacaine 100 mg ketorolac 30 mg epinephrine 400 mcg add Normal saline solution(NSS) to 80 ml divided to two syringes for bilateral periarticular infiltration
  Interventions: Drug: bupivacaine 100 mg
- bupivacaine 200 mg (Active Comparator): bupivacaine 200 mg ketorolac 30 mg epinephrine 400 mcg add NSS to 80 ml divided to two syringes for bilateral periarticular infiltration
  Interventions: Procedure: bupivacaine 200 mg

INTERVENTIONS:
Procedure: bupivacaine 200 mg — bupivacaine 200 mg ketorolac 30 mg epinephrine 400 mcg add NSS to 80 ml divided to two syringes for bilateral periarticular infiltration
  Arms: bupivacaine 200 mg
Drug: bupivacaine 100 mg — bupivacaine 100 mg ketorolac 30 mg epinephrine 400 mcg add NSS to 80 ml divided to two syringes for bilateral periarticular infiltration
  Arms: bupivacaine 100 mg

SUMMARY:
To study efficacy of postoperative pain control of different concentrations of bupivacaine for periarticular infiltration, part of multimodal analgesia, in bilateral total knee arthroplasty.

To study plasma concentration of bupivacaine in patient who received spinal anesthesia and single shot bilateral adductor canal block and periarticular infiltration with bupivacaine for safety level.

DETAILED DESCRIPTION:
Adequate postoperative pain control reduce postoperative morbidity, multimodal analgesia techniques is used for achieve this goal. multimodal analgesia for bilateral total knee arthroplasty are peripheral nerve block, periarticular infiltration, NSAIDs, gabapentins and others. patients undergoing bilateral total knee arthroplasty in siriraj hospital receive spinal anesthesia, single shot bilateral adductor canal block and bilateral periarticular infiltration with bupivacaine so patient receive a large dose of bupivacaine. the investigators study the efficacy of postoperative pain of reduced dose of bupivacaine for periarticular infiltration. and study plasma level of bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old
* American society of anesthesiologists physical status classification 1-3
* Undergoing bilateral total knee arthroplasty with spinal anesthesia and single shot bilateral adductor canal block

Exclusion Criteria:

* Allergy to bupivacaine
* Body weight less than 50 kilograms
* Hepatic disease
* Coagulopathy
* Creatinine clearance less than 60 ml/min
* Uncontrolled cerebrovascular disease
* Hematocrit less than 35%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
postoperative pain score | 0-24 hours postoperative
  Numerical rating scale at rest and movement in the first 24 hours postoperatively

SECONDARY OUTCOMES:
plasma bupivacaine level | 40 minutes after 1st articular infiltration, 15,30,45,60,90 minutes after 2nd periarticular infiltratio
  plasma bupivacaine level at 40 minutes after 1st articular infiltration, 15,30,45,60,90 minutes after 2nd periarticular infiltration
postoperative morphine consumption | first 24 hours and 24-48 hours postoperatively
  postoperative morphine consumption at first 24 hours and 24-48 hours postoperatively
ambulation | 48 hours postoperatively
  patient can walk with assistances within 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: sukanya dej-arkom, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dimitris CN, Taylor BC, Mowbray JG, Steensen RN, Gaines ST. Perioperative morbidity and mortality of 2-team simultaneous bilateral total knee arthroplasty. Orthopedics. 2011 Dec 6;34(12):e841-6. doi: 10.3928/01477447-20111021-02. PMID 22146199
- [Background] Mullaji A, Kanna R, Shetty GM, Chavda V, Singh DP. Efficacy of periarticular injection of bupivacaine, fentanyl, and methylprednisolone in total knee arthroplasty:a prospective, randomized trial. J Arthroplasty. 2010 Sep;25(6):851-7. doi: 10.1016/j.arth.2009.09.007. Epub 2009 Dec 21. PMID 20022457
- [Background] Rosenberg PH, Veering BT, Urmey WF. Maximum recommended doses of local anesthetics: a multifactorial concept. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):564-75; discussion 524. doi: 10.1016/j.rapm.2004.08.003. PMID 15635516
- [Background] Lapmahapaisan S, Chinachoti T, Maisat W, Kleebchan N, Chatsiricharoenkul S, Charoencholvanich K, Rungwattanakij P, Sakulpacharoen N, Sri-In J. Plasma concentrations of bupivacaine after spinal anesthesia with single shot femoral nerve block and periarticular injection in total knee arthroplasty. J Med Assoc Thai. 2014 Jul;97(7):724-9. PMID 25265771
- [Background] Andersen LO, Husted H, Otte KS, Kristensen BB, Kehlet H. High-volume infiltration analgesia in total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Acta Anaesthesiol Scand. 2008 Nov;52(10):1331-5. doi: 10.1111/j.1399-6576.2008.01777.x. PMID 19025523
- [Background] Koh IJ, Kang YG, Chang CB, Kwon SK, Seo ES, Seong SC, Kim TK. Additional pain relieving effect of intraoperative periarticular injections after simultaneous bilateral TKA: a randomized, controlled study. Knee Surg Sports Traumatol Arthrosc. 2010 Jul;18(7):916-22. doi: 10.1007/s00167-010-1051-2. Epub 2010 Jan 30. PMID 20119672
- [Background] Wulf H, Gleim M, Schele HA. Plasma concentrations of bupivacaine after lumbar sympathetic block. Anesth Analg. 1994 Nov;79(5):918-20. doi: 10.1213/00000539-199411000-00017. PMID 7978410
- [Background] Lapmahapaisan S, Chinachoti T, Kongpatanakul S, Chatsiricharoenkul S, Tovnich B, Duangkaew W, Pongnarin P, Sakulpacharoen N, Somcharoen W. Plasma concentrations of bupivacaine after spinal anesthesia with single shot femoral nerve block in total knee arthroplasty. J Med Assoc Thai. 2013 Mar;96(3):312-7. PMID 23539934
- [Derived] Dej-Arkom S, Pangthipampai P, Chandranipapongse W, Chatsirichareonkul S, Narkbunnam R, Charoencholvanich K, Tangchittam S, Iamaroon A. Efficacy and safety of different bupivacaine concentrations in periarticular infiltration combined with adductor canal block for bilateral total knee arthroplasty: a randomized controlled trial. Knee Surg Relat Res. 2024 Jan 19;36(1):5. doi: 10.1186/s43019-024-00211-y. PMID 38243272